CLINICAL TRIAL: NCT01308450
Title: Adult Normative Performance on Quotient ADHD System - Adolescent and Adult Version (Ages 15-55 Years Old)
Brief Title: Adult Normative Performance of the Quotient ADHD System
Acronym: ADHD
Status: Completed | Type: Observational
Sponsor: BioBehavioral Diagnostics Company (Industry)
Responsible Party: Sponsor
Other Study IDs: BBD0111; BBD0111 (Other: BioBehavioral Diagnostics Company)
Record Dates: First submitted 2011-03-02; First posted 2011-03-04 (Estimated); Results first posted 2013-10-30 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: ADHD
Keywords: ADHD Normative Control Group
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Arm, Non ADHD Control Group: Single site, single visit study. Subjects will be administered Standard Rating Scales (Defined) and the Quotient ADHD System Test (Adolescent and Adult Version). Subject's assessed to be Non-ADHD will be eligible to have their Quotient tests added to the Quotient Adolescent and Adult Normative Database.

SUMMARY:
This study is being conducted to enhance and extend the clinical utility of the Quotient® ADHD System Adolescent and Adult Version Test by adding large numbers of well-screened controls to the existing Quotient® ADHD System database of adolescents and adults (ages 15-55).

DETAILED DESCRIPTION:
This study consists of one study visit. Subjects will be recruited using the clinic's relevant patient population. A "Study Recruitment Flyer" will also be posted in various clinic locations (Attachment BBD0111-1). Interested volunteers will participate in an initial screening, which may be done by telephone or in person that will be conducted by the clinic's research staff. Upon preliminary confirmation that the subject meets all inclusion criteria and does not meet any exclusion criteria, an appointment will be scheduled for the study visit.

At the study visit, study will be explained in detail. Adults will be asked to provide written informed consent, parents/guardians of individuals <18 year old will provide written informed consent and minor individual's will provide written assent, prior to any study procedure being performed.

Following consent, a medical history, including current medications the subject is taking, will be obtained. Subjects will complete standard self assessment questionnaires to screen for presence of mental health issues including ADHD, anxiety disorder, depressive disorder or bipolar disorder using the ADHD Self Rating Scale (ASRS), Zung Self-Rated Anxiety Scale (SAS), Zung Self-Rated Depression Scale (SDS), and Mood Disorder Questionnaire (MDQ).

Subjects will not be excluded from the study based on responses to the mental health questionnaires, but results will be considered in the analysis of results.

The subjects will take the 20-minute Quotient® ADHD System Test for Adolescent and Adult assessment.

Subject's assessed to be Non-ADHD will be eligible to have their Quotient tests added to the Quotient Adolescent and Adult Normative Database.

Study Enrollment:

200 Normal control subjects with oversampling of 10%. Total enrollment is expected to be 220.

Study Population:

Male and female subjects from age 15 through 55 years of age. Optimally, there will be approximately 25 subjects per age and gender category but enrollment will not be restricted or limited to these desired categorical goals.

Age Ranges Males Females 15-25 25 25 26-35 25 25 36-45 25 25 46-55 25 25

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for enrollment if they fulfill the following inclusion criteria:

1. Male or Female
2. Ages 15 to 55
3. Un-medicated with medications known to affect ADHD or cognitive functioning
4. Report of good physical health
5. Able to understand test instructions and comply with testing
6. Willing to give written informed consent and/or assent

Exclusion Criteria:

1. History of diagnosis of ADHD
2. History of known neurological disease or insult (e.g., head trauma with LOC, skull fracture, past or present migraine headaches, seizure disorders)
3. Major Medical Disorders
4. Past/present alcohol or substance abuse or dependence
5. Current or past DSM-IV disorder, screened by the computerized SCID I & II, and reviewed by investigator
6. Any major medical or neurological condition that could affect motor activity or attention (e.g. Parkinson's, MS, dementia)
7. Currently ill with cold/flu/infections which may compromise their ability to perform the computer task

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Well-screened, Healthy Non-ADHD Controls, Ages 15-55 from a single private practice clinic.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Focus Center, Clinton, Utah, United States

REFERENCES:
- [Derived] Pivonello R, Muscogiuri G, Holder G, Paul M, Sarp S, Lesogor A, Jordaan P, Eisinger J, Colao A. Long-term safety of long-acting octreotide in patients with diabetic retinopathy: results of pooled data from 2 randomized, double-blind, placebo-controlled phase 3 studies. Endocrine. 2018 Apr;60(1):65-72. doi: 10.1007/s12020-017-1448-5. Epub 2017 Nov 7. PMID 29116540

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 302 subjects meeting enrollment criteria were recruited for this study from a database of patients from a single site, The Focus Center. 300 subjects were eligible to participated and signed Informed Consent.
Pre-assignment Details: This one visit, one site study was conducted to enhance and extend the current "normative" database of the adolescent and adult version of the Quotient ADHD System, an FDA cleared medical device. The study enrolled both male and females, between the ages of 15 and 55 (to match the current database)who were considered "normal", non-ADHD subjects.
Groups:
- Adolescent and Adult Normative Group: Males and Females from ages 15 -55 divided into 4 age groups: 15-25; 26-35;36-45 and 46-55 with each group having approximately equal representation of both genders. Subjects will be recruited to represent a "normative" adolescent and adult sampling of subjects who are not known to have ADHD.
Period: Overall Study
Arm/Group | Adolescent and Adult Normative Group
Started | 302 (302 subjects were screen. 300 subjects were enrolled in this one site, one visit study.)
Completed | 300 (Last subject was enrolled 06/28/2011)
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Adolescent and Adult Normative Group
Number analyzed (Participants) | 302
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22
  Between 18 and 65 years | 280
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 155
  Male | 147
Region of Enrollment [Number; unit: participants]
  United States | 302

OUTCOME MEASURES:

1. Primary Outcome: Well-screened, Non-ADHD Controls to Augment the Existing Adolescent and Adult Database Thus Expanding the Normative Reference Range of Performance of the Quotient® Adolescent and Adult Version Test.
Description: To increase the number of "normal" Adolescent and Adult tests to the existing Quotient System Database. To assure subjects are "normal", participants will complete a standard battery of self assessment questionnaires to screen for the presence of mental health issues including: ADHD, Anxiety Disorder, Depressive Disorder or Bipolar Disorder using the following well established scales and their scoring guidelines:
  1. ADHD Self Rating Scale (ASRS)
  2. Zung Self-Rated Anxiety Scale (SAS)
  3. Zung Self-Rated Depression Scale (SDS)
  4. Mood Disorder Questionnaire (MDQ)
  5. Quotient® ADHD System Test, Adolescent and version Each subject and their individual assessment scores will be evaluated by a physician. Those participants evaluated as "normal"(without ADHD) will have the results of their Quotient test added to the existing Quotient normative database of Non ADHD subjects.
Time Frame: 12 to 18 weeks
Measure: Number; unit: participants
Arm/Group | Adolescent and Adult Normative Group
Number analyzed (Participants) | 300
participants | 300 (300)

ADVERSE EVENTS:
Arm/Group | Adolescent and Adult Normative Group
Serious Adverse Events (participants affected / at risk) | 0/300
Other Adverse Events (participants affected / at risk) | 0/300

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No